CLINICAL TRIAL: NCT02315664
Title: Improving Physical Activity Using an Online Monitoring Tool: a New Model of Care for Knee Osteoarthritis
Brief Title: MONITOR-OA: Using Wearable Activity Trackers to Improve Physical Activity in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Simon Fraser University (Other); Arthritis Research Centre of Canada (Other); Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: H14-01762
Record Dates: First submitted 2014-11-17; First posted 2014-12-12 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-09

CONDITIONS: Knee Osteoarthritis; Joint Diseases
Keywords: Physical activity; Exercise; Osteoarthritis; Knee; Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Motor Activity; Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Intervention Group (Experimental): Education session, Fitbit Flex, and remote coaching by a PT: These three components of the intervention will be delivered to the participants in Month 1 and 2. At the end of the education session, the PT will help participants set personal activity goals. In Month 1 and 2, participants will use the Fitbit Flex. The PT will review the progress with participants via 20-minute bi-weekly phone calls and progressively modify their activities. In Month 3-6, participants will keep the Fitbit and continue to use it with access to a PT via email as needed. In addition, they will receive a monthly e-newsletter about arthritis research that is not related to physical activity.
  Interventions: Behavioral: Education session, Fitbit Flex, and remote coaching by a PT
- Delayed Intervention Group (Experimental): Same intervention with a 2 month delay: The Delayed Intervention Group (control group) will receive the same monthly e-newsletter in Months 1-2. The full intervention will be initiated in Month 3 with a brief education session, use of Fitbit Flex, and counseling by a physiotherapist. In Month 4, they will continue the intervention without the PT phone calls. Participants will keep the Fitbit for Month 5-6, and have email access to PT as needed.
  Interventions: Behavioral: Same intervention with a 2 month delay

INTERVENTIONS:
Behavioral: Education session, Fitbit Flex, and remote coaching by a PT — Participants will receive a brief education session, use of a commercially available physical activity tracker called Fitbit Flex, and remote counseling by a PT. Intervention will be received immediately.
  Arms: Immediate Intervention Group
Behavioral: Same intervention with a 2 month delay — The Delayed Intervention Group will receive the same intervention as the Immediate Intervention Group, but with a 2 month delay.
  Arms: Delayed Intervention Group

SUMMARY:
Physical activity is an essential first-line treatment for patients with knee osteoarthritis (OA). However, a 2013 systematic review found only 13% met the activity recommendation of 150 minutes or more per week. The primary goal of this randomized controlled trail is to assess the efficacy of a physical activity counseling model, involving a group education session, the use of Fitbit Flex (a wireless physical activity tracking device), and online/telephone coaching by a physiotherapist (PT), to improve physical activity and reduce sedentary time in patients with knee OA. Engaging in regular physical activity can have the additional benefit of improving cognitive functioning.

DETAILED DESCRIPTION:
This project will address the Research Question: Can a non-intrusive physical activity tracking tool, combined with a group education session and advice from a physiotherapist (PT), increase physical activity in patients with knee osteoarthritis (OA)? The investigators focus on knee OA because it is common (affecting 1 in 10) and can be debilitating. Being physically active improves pain, mobility and quality of life; however, less than half of patients are active. Combining the best evidence in OA care and digital technology, the investigators propose a new model of care for improving physical activity in patients with OA. Our primary objective is to determine whether a model involving 1) a group education session, 2) the use of Fitbit Flex, a commercially available physical activity tracker, and 3) remote coaching by a PT can improve physical activity and reduce sedentary time in patients with knee OA. This model of care is in line with the goal of Mary Pack Arthritis Program (MPAP) to optimize activity independence of OA patients with MPAP's available human resources. In this proof-of-concept randomized controlled trial (RCT), the investigators hypothesize that compared to a control group (i.e. the Delayed Intervention group), participants in the Immediate Intervention Group will 1) increase moderate/vigorous physical activity (MVPA), 2) reduce sedentary time, 3) improve in OA disease status, and 4) improve in their self-efficacy of OA management, 4) To examine whether individuals in the Intervention Group will show improved cognitive function over the intervention period compared to the control group, and 5) To examine the pre-intervention factors that predict the degree to which individuals in the Intervention Group increase MVPA and reduce sedentary time.

The investigators will use a mixed-methods approach, involving a RCT and in-depth interviews. The proof-of-concept study will employ a stepped wedge RCT design, whereby the intervention will be sequentially rolled out to participants over a number of time periods. The order in which individuals receive the intervention will be determined at random. The strength of this design is that it can properly address the efficacy question, while avoiding the dilemma of withholding the intervention to some participants, as in a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician confirmed diagnosis of knee osteoarthritis OR are both 1) over 50, and 2) have experienced 4 weeks of pain, aching, or discomfort in or around the knee during the last year (equal to or more than 28 separate or consecutive days).
* Have no previous diagnosis of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, polymyalgia rheumatica, connective tissue diseases, fibromyalgia or gout.
* Have no history of using disease-modifying anti-rheumatic drugs or gout medications.
* Have no prior knee replacement surgery, and not on a waiting list for total knee replacement surgery.
* Have no history of acute injury to the knee in the past 6 months.
* Have not had surgery in the back, hip, knee, foot or ankle joints in the past 12 months.
* Have an email address and daily access to a computer with internet connection.
* Be able to attend a 1.5-hour education session at the Mary Pack Arthritis Centre.
* Be able to attend a 1-hour assessment session at Vancouver General Hospital prior to beginning the study, and again 2 and 4 months later.

In addition, participants may be eligible (not required) to partake in a brain magnetic resonance imaging (MRI) assessment if they:

* Do not have a pacemaker, brain aneurysm clip, cochlear implant, electrical stimulator for nerves or bones, implanted infusion pump, artificial heart valve, orthopaedic hardware, other metallic prostheses, coil, catheter or filter in any blood vessel, ear or eye implant, bullets or other metallic fragments.
* Do not have a history of any eye injury involving metal fragments.
* Do not have a history of claustrophobia (i.e. fearful of being in closed or narrow spaces).
* Have not had surgery or tattoos within the past 6 weeks.
* Are able to attend a 1-hour session at the UBC 3T Magnetic Resonance Imaging Centre (2221 Wesbrook Mall, Vancouver).

Exclusion Criteria:

* Have a body mass index of equal to or greater than 40
* Have received a steroid injection in a knee in the last 6 months
* Have received a hyaluronate injection in a knee in the last 6 months
* Use medication that may impair activity tolerance (e.g. beta blockers)
* Are at risk when exercising, as identified by the Physical Activity Readiness Questionnaire (PAR-Q)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — Arthritis Research Canada
Locations (1):
- Arthritis Research Canada, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falck RS, Best JR, Li LC, Chan PCY, Feehan LM, Liu-Ambrose T. Can we improve cognitive function among adults with osteoarthritis by increasing moderate-to-vigorous physical activity and reducing sedentary behaviour? Secondary analysis of the MONITOR-OA study. BMC Musculoskelet Disord. 2018 Dec 21;19(1):447. doi: 10.1186/s12891-018-2369-z. PMID 30577819
- [Derived] Li LC, Sayre EC, Xie H, Falck RS, Best JR, Liu-Ambrose T, Grewal N, Hoens AM, Noonan G, Feehan LM. Efficacy of a Community-Based Technology-Enabled Physical Activity Counseling Program for People With Knee Osteoarthritis: Proof-of-Concept Study. J Med Internet Res. 2018 Apr 30;20(4):e159. doi: 10.2196/jmir.8514. PMID 29712630
- See also: Study webpage — http://arthritis.rehab.med.ubc.ca/2015/03/03/improving-physical-activity-using-an-online-monitoring-tool-a-new-model-of-care-for-knee-osteoarthritis-monitor-oa/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from February 2015 - October 2016. Recruitment strategies included placing study advertisement material at Community Health Centres and Mary Pack Arthritis Centre. We also had study advertisement disseminated through Arthritis Research Canada website and group collaborators' group newsletters.
Pre-assignment Details: After enrollment, participants completed the baseline assessment, and after completion of baseline participants were randomly assigned to the immediate group or the delayed group (ie, control) in 1:1 allocation ratio.
Period: Overall Study
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Started | 30 | 31
Completed | 29 | 27
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Group | Delayed Intervention Group | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.4) | 62.1 (8.5) | 61.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 8 | 3 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 31 | 61
Marital Status [Count of Participants; unit: Participants]
  Married/Common Law | 19 | 14 | 33
  Separated/Divorced | 7 | 8 | 15
  Widowed/Never married/Other | 4 | 9 | 13
Gross annual household income (CAN$) [Count of Participants; unit: Participants]
  ≤12,000 | 0 | 0 | 0
  12,001-24,000 | 1 | 2 | 3
  24,001-40,000 | 4 | 2 | 6
  40,001-60,000 | 5 | 6 | 11
  60,001-80,000 | 9 | 4 | 13
  80,001-100,000 | 2 | 3 | 5
  >100,000 | 5 | 6 | 11
  No answer | 4 | 8 | 12
Diagnosed with OA [Count of Participants; unit: Participants]
  Yes | 26 | 26 | 52
  No, but met the "likely OA" criteria | 4 | 5 | 9
In general would you say your health is... [Count of Participants; unit: Participants]
  Excellent | 1 | 0 | 1
  Very good | 15 | 14 | 29
  Good | 10 | 14 | 24
  Fair | 4 | 3 | 7
  Poor | 0 | 0 | 0
Compared to one year ago, how would you rate your health in general now? [Count of Participants; unit: Participants]
  Much better | 2 | 2 | 4
  Somewhat better | 6 | 3 | 9
  About the same | 12 | 15 | 27
  Somewhat worse | 10 | 11 | 21
  Much worse | 0 | 0 | 0
Number of comorbid conditions [Median (Inter-Quartile Range); unit: Comorbid conditions] | 2.0 [1.0 to 4.0] | 4.0 [2.0 to 5.0] | 3.0 [2.0 to 4.0]
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (5.5) | 29.2 (4.8) | 29.2 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Moderate-to-Vigorous Physical Activity (MVPA)
Description: Participants wore a SenseWear Mini accelerometer for 7 days at baseline, and Months 2, 4, and 6. We calculated the average daily time (minutes) spent in MVPA accumulated in bouts. A bout is defined as 10 or more consecutive minutes at the level of 3 or higher METs, with allowance for interruption of up to 1 minute below the threshold.
Time Frame: Baseline; 2 months, 4 months and 6 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: Minutes per day
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
Minutes per day
  Baseline | 62.1 (54.6) | 65.3 (77.4)
  2 months | 75.5 (54.3) | 50.0 (46.8)
  4 months | 62.6 (56.3) | 60.1 (76.8)
  6 months | 65.6 (48.5) | 70.7 (71.9)

2. Secondary Outcome: Time Spent in Sedentary Behaviors
Description: We calculated the average daily time spent with an energy expenditure of 1.5 METs or lower, occurring in bouts of 20 minutes or more during waking hours.
Time Frame: Change from baseline in time spent sedentary behaviors at 2 months, 4 months, and 6 months.
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: Minutes per day
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
Minutes per day
  Baseline | 464.1 (137.7) | 497.4 (200.7)
  2 months | 437.6 (133.9) | 503.0 (160.7)
  4 months | 505.9 (167.2) | 508.9 (189)
  6 months | 435.8 (138.8) | 496.0 (179.5)

3. Secondary Outcome: KOOS - Symptoms
Description: Symptoms were measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 2 months, 4 months and 6 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
score on a scale
  Baseline | 59.8 (16.1) | 62.9 (17.2)
  2 months | 62.6 (15.6) | 61.7 (14.5)
  4 months | 62.4 (14.7) | 63.4 (16.7)
  6 months | 62.1 (15.3) | 61.4 (19.8)

4. Secondary Outcome: KOOS - Pain
Description: Pain was measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 2 months, 4 months and 6 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
score on a scale
  Baseline | 66.2 (17.5) | 65.1 (17.9)
  2 months | 70.9 (17) | 64.8 (14.6)
  4 months | 67.5 (15.5) | 66.3 (15.2)
  6 months | 68.6 (17.5) | 66.2 (16.4)

5. Secondary Outcome: KOOS - Activity of Daily Living
Description: Activity of Daily Living was measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 2 months, 4 months and 6 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
score on a scale
  Baseline | 71.8 (17.5) | 74.1 (17.6)
  2 months | 76 (16.1) | 71 (16.5)
  4 months | 76.6 (17.5) | 75.2 (17.2)
  6 months | 75.1 (15.9) | 73.9 (15.8)

6. Secondary Outcome: KOOS - Sports & Recreation
Description: Sports & Recreation was measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 2 months, 4 months and 6 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
score on a scale
  Baseline | 47.3 (26.6) | 52.7 (27.7)
  2 months | 49.3 (24.9) | 47 (23.3)
  4 months | 50 (25.6) | 48.9 (27.7)
  6 months | 50.4 (26.3) | 49.8 (29.2)

7. Secondary Outcome: KOOS - Quality of Life
Description: Quality of Life was measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 2 months, 4 months and 6 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
score on a scale
  Baseline | 41 (19.8) | 44.6 (16.3)
  2 months | 47.2 (18.9) | 42.4 (16.8)
  4 months | 45.4 (17.6) | 47.5 (13.6)
  6 months | 44.9 (17.9) | 48.1 (19.1)

8. Secondary Outcome: Partners in Health Scale
Description: The Partners in Health Scale is a 12-item measure designed to assess self-efficacy, knowledge of health conditions and treatment, and self-management behaviors such as adopting a healthy lifestyle. Scores range from 0 to 96, with lower being better.
Time Frame: Baseline; 2 months, 4 months and 6 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 30 | 31
score on a scale
  Baseline | 18.4 (12.6) | 20.5 (12.8)
  2 months | 14.9 (11.4) | 18.3 (13.7)
  4 months | 14.3 (10.1) | 14.9 (9.6)
  6 months | 12.9 (9.2) | 13.1 (9.2)

ADVERSE EVENTS:
Time Frame: During the data collection for the randomized controlled trial, adverse event data was tracked using a monthly log (self-reported) by the participant.
Description: We tracked self-reported adverse events (falls, cardiovascular and musculoskeletal events).
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

LIMITATIONS AND CAVEATS:
Our sample was relatively active; hence, the results may not be generalizable to people with knee OA who are more sedentary. Also, the long-term effect of the intervention remained unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02315664/Prot_SAP_000.pdf